CLINICAL TRIAL: NCT05222061
Title: A ProSpecTivE, RaNdomIzed Trial of Drug Coated Balloon For tReating the Side
Brief Title: A Study of Drug Coated Balloon For Treating the Side Branch in Complex Bifurcation Lesions
Acronym: STENT-FREE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Dmitrii Khelimskii, MD, PhD, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-45
Record Dates: First submitted 2021-04-15; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug coated balloon, coronary bifurcation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- provisional-stenting group (Active Comparator): Provisional stenting will be performed according to european bifurcation club consensus. MB and SB predilatation will be at the operator's discretion. A stent is delivered in the main vessel and positioned across the bifurcation. POT is mandatotary. In case of dissection impeding the flow in the SB or acute coronary closure after MB atenting a SB stenting using a DES was allowed. Dual-stent techniques will be performed according to the recommendation of the EBC consensus.
  Interventions: Device: Conventional balloon for the side brunch
- DCB group (Experimental): Coronary guidewires should be passed to the MB and SB, respectively. Lesion preparation of the main branch should be undertaken as considered necessary. Lesion preparation of the side branch is mandatorary. If the angiographic result will be good after predilatation (residual stenosis < 30%), drug-eluting stent will implanted in the main branch of the bifurcation site (the stent diameter should be choosen based on the diameter of the distal MB). A kissing with conventional balloons should be performed in the MB and SB. Reapet kissing with drug-coated balloonin the SB and conventional balloon in MB (30 seconds at low pressure (8-10 bar) should be performed. The DCB diameter was again 0.8-1.0 of the vessel diameter.
  In case of dissection impeding the flow in the SB or acute coronary closure after DCB application a SB stenting using a DES was allowed. Dual-stent techniques will be performed according to the recommendation of the EBC consensus.
  Interventions: Device: Drug coated balloon for the side brunch

INTERVENTIONS:
Device: Drug coated balloon for the side brunch — Intervention is explained in group description
  Arms: DCB group
Device: Conventional balloon for the side brunch — Intervention is explained in group description
  Arms: provisional-stenting group

SUMMARY:
Hypothesis: In patients undergoing coronary stenting for the true bifurcation lesions, main branch stenting followed by side branch dilatation with drug coated balloon is superior to the provisional-stenting strategy in terms of late lumen loss at 12 months.

DETAILED DESCRIPTION:
Although drug-eluting stents are still the default interventional treatment of coronary artery disease, drug-coated balloons (DCBs) represent an alternative therapeutic strategy in certain anatomic conditions. Although their use is established for in-stent restenosis of both bare-metal and drug-eluting stents, recent clinical data demonstrate promising results in de novo small-vessel disease, myocardial infarction and bifurcation settings.

Patients with coronary bifurcation lesions account for approximately 15% to 20% of all coronary lesions in coronary interventional procedures. Despite the use of drug-eluting stents, treating bifurcation lesions remains challenging especially in settings of side branch involvment. PCI of such lesions is associated with lower immediate angiographic and clinical success and higher rates of restenosis, which, in addition, are more challenging to treat compared to non-bifurcated lesions.

The optimal treatment of patients with biffurcations lesions involving SB is as yet undefined. Despite provisional stenting strategy is the preferred technique for most patients. Several studies demonstrated that two-stent techniques may be preferable in patients with true bifurcation lesions. However, as a general approach, the EBC suggests conducting PCI procedures with the aim of limiting the amount of stent metal implanted.

In this settings the use of DCB for bifurcation lesions may have some advantages. DCB provides a smaller profile compared with DES, allowing better SB access. The lack of foreign body implantation with DCB obviates the risk for stent thrombosis and may allow for a shorter duration of dual-antiplatelet therapy compared with DES.

To date, there have been very few clinical trials on the treatment of bifurcation lesions with drug-eluting balloons and all of these included only a small cohort of patients.

Early studies looking into the use of a BMS in the MB in combination with a DCB in the SB demonstrated a low late lumen loss in the SB when treated alone with a DCB [9]; recent observational studies focusing largely on a SB DCB combined with an MB DES strategy showed good SB results.

In the register PEPCAD V, 28 patients with lesions involving coronary bifurcation were treated by DCB Sequent Please in the secondary branch and the main vessel, BMS implantation in the main vessel, opening the stent struts toward the SD with only one balloon. At 9 months, the LLL in the MB was 0.38 ± 0.46 and 0.21 ± 0.48 mm in the SB resulting in an MLD of 2.2 ± 0.60 mm in the MB and 1.7 ± 0.44 mm in the SB. Three patients had angiographic restenosis, and in one a TLR was performed. Two patients experienced a late stent thrombosis at 6 and 8 months.

Improvement in the technique of intervention with the use of DES and DCB was observed in the prospective multicenter, non-randomized study DEBSIDE. Data from 50 patients were included,. Predilatation of both branches was performed with conventional balloons, then provisional stenting of MB using DES, kissing dilatation with conventional balloons. Authors proposed to remove guidewire from the MB in order to reduce the friction of the DCB and the loss of the antiproliferative drug from the surface of the balloon when it was delivered to the SB, to inflate the balloon with a pressure of 8-10 atmospheres for 30 seconds. Coronary angiography after 6 months, showed the LLL in the SB was 0.04 ± 0.34 mm, and in the MB, 0.54 ± 0.60 mm. The revascularization rate at 12 months was 6% and 2% in MB and SB, respectively.

A prospective multicenter study by Iannopollo G. analyzed results of the Agent DCB application in the real-world population. Among the 354 patients included in the registry (450 lesions treated with 508 DCBs), DCBs were used for the treatment of bifurcation lesions in 26%. DCB was inflated in the SB with a pressure of 8 atmospheres for 60 seconds after provisional stenting of the MB with the DES. The frequency of MACE after 544 days was 3.7%.

In the case of restenosis, DCB considered today a valuable alternative to DES, with strong evidence for the treatment of both BMS and DES restenosis. With its advantage of avoiding the creation of a dual stent layer in the coronary arteries, their use seems particularly attractive especially in patients with complex bifurcation lesions. In these settings DCB does seem to be a promising strategy, however, large randomised clinical trials are needed to show the safety and efficacy of this technology.

ELIGIBILITY:
Inclusion Criteria:

* Main branch and side branch diameter both >2.5 mm, evaluated based on coronary angiography, performed no later than 6 month before baseline visit;
* Patient ≥18 years old;
* Signed informed consent;
* True bifurcation lesion type 1:1:1 or 0:1:1 or 1:0:1 and
* ischemic symptoms, or
* positive non-invasive imaging for ischemia, or
* positive fractional flow reserve

Exclusion Criteria:

1. ST Elevation Miocardial Infarction <72 hours preceding;
2. Cardiogenic shock;
3. Chronic total occlusion of either main or side branch of the bifurcation;
4. >2 other coronary lesions planned for treatment;
5. SYNTAX score >32;
6. Left main stenosis;
7. In-stent restenosis;
8. Renal function insufficiency: Serum creatinine > 177 mmol/l; or undergoing hemodialysis;
9. Left ventricular ejection fraction ≤ 30%;
10. Patient life expectancy less than 12 months;
11. Patient's inability to fully cooperate with the study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss for both main branch and side branch | 12 months
  Measured by quantitative coronary angiography.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 3,6,12 months
  Includes cardiac death, myocardial infarction in target vessel territory, clinically Indicated target lesion revascularization
All-cause death | 3,6,12 months
Stent/vessel thrombosis | 3,6,12 months
  According to the definition of ARC (definite or probable)
Angiographic Binary Restenosis | 12 months
  Measured by quantitative coronary angiography.
Target Lesion Revascularization | 3,6,12 months
  TLR is defined as any ischemia-driven repeat PCI of the target lesion (including 5 mm proximal and distal to the target lesion) or bypass surgery of the target vessel.
Target Vessel Revascularization | 3,6,12 months
  TVR as any ischemia-driven repeat PCI or bypass surgery of the target vessel. The target vessel consists of target lesion(s) and any additional lesions in the main epicardial coronary artery or branches containing the target lesion.
Angina status | 3,6,12 months
  Change in the stable angina functional class according to Canadian Cardiovascular Society
Angiographic success in main branch and side branch | immediately after the procedure
  Defined as a residual stenosis <30% and TIMI flow grade 3 at the end of the procedure in the MB and SB respectively
Fluoroscopic time | immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin National Medical Research Center, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No